CLINICAL TRIAL: NCT03672812
Title: Randomized Clinical Trial to Evaluate the Use of Liraglutide in Individuals With Brain Death and Anti-inflammatory and Anti-apoptotic Effects on Organs to be Transplanted
Brief Title: The Use of Liraglutide in Brain Death
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 87650318100005327
Record Dates: First submitted 2018-09-13; First posted 2018-09-17 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Brain Death
Keywords: liraglutide; brain death; inflammation
MeSH Terms: conditions — Brain Death; Inflammation | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo (No Intervention): 0,5ml
- liraglutide (Experimental): 0,5ml
  Interventions: Drug: Liraglutide

INTERVENTIONS:
Drug: Liraglutide — liraglutide 3mg 6/6 hours
  Other Names: placebo
  Arms: liraglutide

SUMMARY:
There is evidence of the association of brain death and inflammation, affecting outcomes of transplanted organs, but in a way not fully understood. Observational studies suggest that the use of target-guided therapies has a beneficial effect in reducing the rate of donor loss due to cardiac arrest and increasing the rate of donor-picked organs, which will be tested through the randomized clinical trial. However, no study so far has directly tested the effect of drugs with anti-inflammatory and anti-apoptotic properties administered to the donor in encephalic death in reducing inflammation of organs to be transplanted. This study aims to evaluate the use of liraglutide in patients with brain death in relation to their ability to attenuate the inflammation induced by encephalic death by means of a randomized clinical trial.

DETAILED DESCRIPTION:
The intervention group will be composed of individuals deceased in brain dead, after the conclusion of the brain dead protocol by the teams responsible for the Intensive care and will receive liraglutide. The control group will be composed of the same population of individuals who died in brain dead of the intervention group, but will receive a placebo.

ELIGIBILITY:
Inclusion Criteria:

* individuals deceased more than 18 years after the end of the brain death protocol

Exclusion Criteria:

* Pregnant women, patients with advanced renal failure on hemodialysis, with hepatic insufficiency or allergy known to liraglutide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
change inflammation | from 6 hours to 24 hours
  change interleukin 6

SECONDARY OUTCOMES:
change inflammation with liraglutide | from 6 to 24 hours
  change interleukin 8
change inflammation liraglutide group | from 6 to 24 hours
  change interleukin 10
change inflammation intervention group | from 6 to 24 hours
  change tumor necrosis factor-alpha
change inflammation | from 6 to 24 hours
  change interferon gamma

CONTACTS AND LOCATIONS:
Overall Officials: Cristiane Leitao, PhD, Principal Investigator — Hospital de Clinicas de Porto Alegre
Locations (1):
- Hospital Santa Isabel, Blumenau, Santa Catarina, Brazil

IPD SHARING:
Plan to Share IPD: Undecided